CLINICAL TRIAL: NCT00188851
Title: A Prospective Randomized Trial of Structured Treatment Interruption(STI) Followed by Initiation of a New Antiretroviral Regimen(ARV) Versus Immediate Switching to a New ARV in HIV-Infected Patients Experiencing Virologic Failure on HAART
Brief Title: Structured Treatment Interruption for HIV Patients With Virologic Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); CIHR Canadian HIV Trials Network (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIHR82716
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: HIV
Keywords: HIV; salvage regimen; virologic failure; treatment interruption; ARV experienced

INTERVENTIONS:
Drug: therapeutic management strategy

SUMMARY:
The purpose of this study is to assess the virologic impact of switching treatment-experienced HIV-infected patients with virologic failure to a salvage regimen with or without a 12 week STI prior to the switch.

Hypothesis: A STI prior to starting a salvage regimen will result in an improved virologic response.

DETAILED DESCRIPTION:
To prospectively determine the virologic impact of switching treatment-experienced HIV-infected patients with virologic failure to a salvage regimen with or without a 12 week STI prior to the switch.

Hypothesis: By withdrawing ARV drug pressure, resistant HIV virus will revert to wild-type. In treatment-experienced HIV patients who experience virologic failure, a STI prior to starting a salvage regimen will result in an improved virologic response and more prolonged vral suppression compared to immediate switching to a new regime.

Interventions:

Immediate Switch to Salvage Therapy: Patients randomized to the control arm will be switched immediately to a salvage regimen using the information from the treatment history and genotype results.

Structured Treatment Interruption: Patients randomized to the STI arm will have their present regimen stopped for 12 weeks and will have a genotype repeated in the 12th week. A salvage regimen will be started at week 12 using the information from the treatment history and baseline genotype results.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* On therapy with a triple ARV that includes a protease inhibitor and/or non-nucleoside reverse transcriptase inhibitor for the past 3 months with no changes in any agent of the combination in the past 14 days.
* Virologic failure while on the combination as defined by a plasma HIV RNA > 1000 copies/mL measured on 2 occasions at least 4 weeks apart.
* HIV RNA <500,000 copies/mL.
* CD4 cell count must be > 50/mm3
* Patients must not have a present history of opportunistic infections or acute illness requiring treatment within the preceding 30 days.
* The patient has at least two new ARV available based on history, and at least two of these new agents will be included in the new salvage regimen.

Exclusion Criteria:

* Active substance abuse which would interfere with the patient's ability to participate in this trial, or declared non-compliance.
* Pregnancy or breast feeding.
* Patients with any of the following abnormal laboratory test results at screening:· Hemoglobin<80 g/L, neutrophil count<750 cells/mL, Platelet<20,000 /mL· AST or ALT > 5X Upper Limit of Normal (ULN)· Creatinine > 250 umol/L
* End stage organ disease
* Patient with malignancy receiving systemic chemotherapy
* Patient has need for immune modulators (interleukin, interferon, GMCSF etc) or prednisone. This excludes a short course of inhaled or oral steroids for asthma exacerbation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196
Dates: Start 2001-01; Study Completion 2005-11

PRIMARY OUTCOMES:
To prospectively determine the virologic impact of switching treatment-experienced HIV-infected patients with virologic failure to a salvage regimen with or without a 12 week STI prior to the switch.

SECONDARY OUTCOMES:
1. To prospectively determine differences in other virologic parameters through follow up between patients being switched to a salvage regimen with or without a STI.
2. To prospectively determine differences in change in CD4 count through follow up and at 24, 48 and 60 weeks following randomization between patients being switched to a salvage regimen with or without a STI.
3. To prospectively determine differences in the development or reactivation of opportunistic infections and survival between patients being switched to a salvage regimen with or without a STI at 60 weeks following randomization
4. To determine the proportion of virus of patients being treated with a STI that converts to wild-type and how that relates to the virologic response (% of patients with undetectable viral load sustained for 3 months).
5. To determine the impact of the STI on quality of life measures.
6. To determine the genotypic resistance pattern of virus from patients who fail treatment after suppression to <50 copies/mL on the salvage regimen and to compare results in those who do and do not receive an STI.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Loutfy, MD, Study Chair — University Health Network, Toronto, On; Joel Singer, MD, Study Director — Canadian Trials Network, Vancouver, B.C.; Janet Raboud, Dr., Study Director — Univeristy Health Network, Toronto, On; Stephen Shafran, MD, Study Director — University of Alberta, Edmonton, Alberta; Bill Cameron, MD, Study Director — Ottawa Hospital, Ottawa, On; Sylvie Trottier, MD, Study Director — Clinique Medicale L'Actuel, Montreal, Quebec; Richard Harrigan, MD, Study Director — B.C. Centre of Excellence, Vancouver, B.C.